CLINICAL TRIAL: NCT03660527
Title: Nutritional Status of Residents From the Chinese National Health and Nutrition Survey During 2010-2012
Brief Title: Nutritional Status of Chinese Residents
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Principal Investigator, Lichen Yang, National Institute for Nutrition and Health, Centers for Disease Control and Prevention, China
Other Study IDs: Nutrition survey
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Nutrition Status of Chinese Residents
Keywords: hemoglobin, vitamin D, vitamin A, TC, TG, HDLC

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 6-17 year old
  Interventions: Other: Not refered
- 18-44 year old
  Interventions: Other: Not refered
- 45-59 year old
  Interventions: Other: Not refered
- above 60 year old
  Interventions: Other: Not refered

INTERVENTIONS:
Other: Not refered — No intervention was refered.

SUMMARY:
In this study, we analyzed the nutritional status of Chinese residents aged above 6y. The indicators such as the hemoglobin, vitamin D, vitamin A and TG, TC and HDLC were also included. Related risk factors (such as age, region type, ethnicity, bodyweight, height, education, season, smoke habit, etc).

ELIGIBILITY:
Inclusion Criteria:

* Participanted in China national nutrition and health survey (CNNHS) 2010-2012; Aged above 6 years old; Had blood taken;

Exclusion Criteria:

* No.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participanted in China national nutrition and health survey (CNNHS) 2010-2012; Aged above 6 years old; Had blood taken;
  Exclusion Criteria:
Sampling Method: Probability Sample
Enrollment: 41420 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2013-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
anemia status | through study completion, an average of 1 year
vitamin D deficiency | through study completion, an average of 1 year
vitamin A deficiency | through study completion, an average of 1 year
Metabolic syndrome | through study completion, an average of 1 year

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282